CLINICAL TRIAL: NCT02240628
Title: In Children, Placing a Synera Patch for Intravenous Access Combined With Administration of a Propofol-Lidocaine Mixture Decreases Pain Associated With Propofol Intravenous Injection.
Brief Title: Combining Placing a Synera Patch With Propofol/Lidocaine Mixture to Decrease Pain With IV Propofol Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor Of Pediatric Anesthesia, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-14-0323
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Pain on IV Injection of Propofol.
MeSH Terms: interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol-Lidocaine mixture (Active Comparator): All patients from both groups will receive a Synera Patch. Patients in this group will receive Propofol mixed with Lidocaine. Pain will be evaluated during the Propofol injection by both a blinded observer and a blinded anesthesia member.
  Interventions: Device: Lidocaine/tetracaine transdermal patch; Drug: Lidocaine
- Propofol -Saline mixture (Placebo Comparator): All patients from both groups will receive a Synera Patch. Patienst in this group will receive Propofol mixed with Saline. Pain will be evaluated on Propofol injection by both a blinded observer and a blinded anesthesia member.
  Interventions: Device: Lidocaine/tetracaine transdermal patch; Drug: Saline

INTERVENTIONS:
Device: Lidocaine/tetracaine transdermal patch — All patients in arm 1 and arm 2 will receive the Synera Patch.
  Other Names: NDC 43469-864-01; Synera Patch
Drug: Saline — Patients in arm 2 will receive Saline with the Propofol.
  Other Names: 0.9% sodium chloride solution.
  Arms: Propofol -Saline mixture
Drug: Lidocaine — Patients in arm 1 will receive Lidocaine with the Propofol.
  Arms: Propofol-Lidocaine mixture

SUMMARY:
The main objective is to evaluate if combining placing the Synera patch and using Propofol /Lidocaine mixture will further decrease the pain associated with the IV injection of Propofol.

DETAILED DESCRIPTION:
Commonly, anesthesiologists inject Propofol, a sleeping medication, intravenously to induce general anesthesia.Propofol injection is commonly associated with burning pain. In a previous onsite study we concluded that placing a Synera patch at least 30 minutes before placing the IV decreased the pain associated with the Propofol injection. Also,a study documented that adding Lidocaine to the Propofol decreases the pain associated with propofol injection. In our study here we are trying to evaluate if combining the use of both the Synera patch and the Propofol-Lidocaine mixture will further decrease the pain associated with the IV Propofol injection.

All children will receive a Synera Patch, it will be placed on the dorsum of both hands for at least 30 minutes.All Children will be Sedated with P.O Versed.

22 g IV will be started either in the holding area or in the OR. Children will be randomized into groups using a computer generated randomization list:- Group 1 will receive Propofol -Lidocaine mixture. Group 2 will receive Propofol-Saline mixture. An independent blinded observer and an anesthesia member will independently evaluate pain on Propofol injection according to pain scale.

1. No pain.
2. Mild Pain (associated with facial expression of pain).
3. Moderate Pain(Pulling the arm).
4. Severe Pain (screaming).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children 6-17 yrs.
* Scheduled to receive general anesthesia for an elective procedure.
* ASA classification 1-2

Exclusion Criteria:

* Children with Skin disease and/or Skin infections.
* Allergy to Propofol, Lidocaine or tetracaine.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: samia khalil, M.D, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol-Lidocaine Mixture | Propofol -Saline Mixture
Started | 38 | 38
Completed | 32 | 33
Not Completed | 6 | 5
Not completed — Physician Decision | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol-Lidocaine Mixture | Propofol -Saline Mixture | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3750 (2.2683) | 14.5455 (2.0930) | 14.46025 (2.18065)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Children in Each Group Who Don't Feel Pain or Have Mild Pain on Propofol Injection.
Time Frame: During propofol injection.
Measure: Number; unit: participants
Arm/Group | Propofol-Lidocaine Mixture | Propofol -Saline Mixture
Number analyzed (Participants) | 32 | 33
participants | 29 | 19

2. Secondary Outcome: Pain Intensity
Description: A blinded independent observer will rate pain on Propofol injection according to a pain scale.
  1. No pain.
  2. Mild pain(associated with facial expression of pain).
  3. Moderate Pain(Pulling/withdrawal of arm).
  4. Severe Pain(Screaming).
Time Frame: During Propofol injection.
Measure: Number; unit: participants
Arm/Group | Propofol-Lidocaine Mixture | Propofol -Saline Mixture
Number analyzed (Participants) | 32 | 33
participants
  1 | 20 | 6
  2 | 9 | 13
  3 | 1 | 6
  4 | 2 | 8

ADVERSE EVENTS:
Arm/Group | Propofol-Lidocaine Mixture | Propofol -Saline Mixture
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 2/32 | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Propofol-Lidocaine Mixture (N=32) | Propofol -Saline Mixture (N=33)
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 — Erythema at site of the Synera patch was noted after removal of the patch which resolved by itself.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes